CLINICAL TRIAL: NCT05001802
Title: Transverse Versus Longitudinal Technique of Ultrasound-Guided Transmuscular Quadratus Lumborum Block:A Randomized Controlled Study Comparing Dermatomal Spread
Brief Title: Comparison of Two Techniques of Quadratus Lumborum Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Cui Xulei, associate professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 20210505
Record Dates: First submitted 2021-05-19; First posted 2021-08-12 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Nerve Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transverse quadratus lumborum block (Active Comparator): The patients will receive the transmuscular quadratus lumborum block before surgery using the transverse scan, in-plain, posterior to anterior approach. 0.6ml/kg 0.375% ropivacaine is injected when the correct needle location is confirmed.
  Interventions: Procedure: transverse scan, in-plane, posterior- anterior quadratus lumborum block
- longitudinal quadratus lumborum block (Experimental): The patients will receive the transmuscular quadratus lumborum block before surgery using the paramedic sagittal longitudinal scan, in-plain, caudal-cephalic approach.0.6ml/kg 0.375% ropivacaine is injected when the correct needle location is confirmed.
  Interventions: Procedure: paramedian sagittal longitudinal scan, in-plane, caudal-cranial quadratus lumborum block

INTERVENTIONS:
Procedure: transverse scan, in-plane, posterior- anterior quadratus lumborum block — transverse scan, in-plane, posterior- anterior quadratus lumborum block The patients will receive the transmuscular quadratus lumborum block before surgery using the transverse scan, in-plain, posterior to anterior approach. 0.6ml/kg 0.375% ropivacaine is injected when the correct needle location is confirmed.
  Other Names: drug:ropivacaine
  Arms: transverse quadratus lumborum block
Procedure: paramedian sagittal longitudinal scan, in-plane, caudal-cranial quadratus lumborum block — The patients will receive the transmuscular quadratus lumborum block before surgery using the paramedic sagittal longitudinal scan, in-plain, caudal-cephalic approach.0.6ml/kg 0.375% ropivacaine is injected when the correct needle location is confirmed.
  Other Names: drug:ropivacaine
  Arms: longitudinal quadratus lumborum block

SUMMARY:
Our objective is to investigate the extent of cranial dermatomal spread of transmuscular quadratus lumborum block(TMQLB )when equal dosage(ml/kg) of local anesthetic are injected with the transverse versus an modified paramedian sagittal approach for patients undergoing laparoscopic adrenalectomy.

DETAILED DESCRIPTION:
The paramedian sagittal oblique transmuscular quadratus lumborum block(TMQLB )approach has been introduced to facilitate cranial spread by injecting the local in a caudal to cranial direction compared with the transverse approach. Currently, there are no data comparing the two techniques mentioned above with regards to extent of spread level. Our objective is to investigate the extent of cranial dermatomal spread of TMQLB when equal dosage(ml/kg) of local anesthetic are injected with the transverse versus an modified paramedian sagittal approach for patients undergoing laparoscopic adrenalectomy. In addition, the investigators wish to compare the performance time, caudal dermatomal spread of TMQLB and postoperative analgesia effect.

ELIGIBILITY:
Inclusion Criteria:

* ≥Age 18yrs

  * American Society of Anesthesiologists physical status I-II
  * Undergo laparoscopic adrenalectomy
  * Informed consent
  * Able to cooperate with study process

Exclusion Criteria:

* Allergy to local anesthetic and other medications used in the study
* Patient refusal or lack of informed consent
* Coexisting hematological disorder or with deranged coagulation parameters
* Pre-existing major organ dysfunction such as hepatic and renal failure
* History of previous renal surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-08-20 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Cephalic sensory dermatomal spread | 20 minutes after block performance]
  The pinprick method at the midclavicular line was used to assess the extent of the dermatomal blockade, 20 minutes following the completion of the procedure by a person who was blinded to group allocation. The most cephalic dermatomal level that show a decreased pinprick sensation is recorded.A block failure was defined as the absence of any demonstrable sensory block 20 minutes after performance of the block.

SECONDARY OUTCOMES:
Time to performance of procedure | Duration of procedure
  Duration from needle insertion toward local anesthetic injection finished
Total sensory dermatomal spread | 20 minutes after block performance
  The pinprick method at the midclavicular line was used to assess the extent of the dermatomal blockade, 20 minutes following the completion of the procedure by a person who was blinded to group allocation. The total number of dermatomal levels that show decreased pinprick sensation is recorded.A block failure was defined as the absence of any demonstrable sensory block 20 minutes after performance of the block.
Incidence of complication | Within 48 hours after surgery
  incidence of complication including bleeding, hematoma, infection at puncture site, local anesthetic poisoning, etc
Caudal sensory dermatomal spread | 20 minutes after block performance
  The pinprick method at the midclavicular line was used to assess the extent of the dermatomal blockade, 20 minutes following the completion of the procedure by a person who was blinded to group allocation. The most caudal dermatomal level that show a decreased pinprick sensation is recorded.A block failure was defined as the absence of any demonstrable sensory block 20 minutes after performance of the block.
rescue analgesics usage | At 0,12,24,48 hours after surgery
  NSAIDs or opioids used for pain relief and their dosage

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China